CLINICAL TRIAL: NCT01315431
Title: A Phase I Study of Tesetaxel Administered in Combination With Capecitabine to Subjects With Solid Tumors
Brief Title: A Study of Tesetaxel Plus Capecitabine in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOST107
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumor
Keywords: Solid tumor malignancy, excluding lymphoma
MeSH Terms: interventions — tesetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tesetaxel-capecitabine (Experimental)
  Interventions: Drug: Tesetaxel plus capecitabine

INTERVENTIONS:
Drug: Tesetaxel plus capecitabine — Study medication, which will include tesetaxel capsules and capecitabine tablets, will be administered orally for two 21-day cycles. In each cycle, tesetaxel will be administered at a dose of 27 mg/m2 on Day 1, and capecitabine will be administered in Cohort 1 at a dose of 2000 mg/m2/day and in Cohort 2 at a dose of 1750 mg/m2/day (in 2 equally divided doses) on Day 1 through Day 14.
  At the conclusion of Cycle 2, patients who, in the opinion of the investigator, appear to have benefitted from protocol therapy may receive up to 6 additional cycles under a separate protocol.
  Other Names: DJ-927; Xeloda

SUMMARY:
This study is being performed to confirm the safety of tesetaxel 27 mg/m2 (Day 1) in combination with capecitabine 2000/mg/m2/day (in 2 equally divided doses on Days 1 through 14) in a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Confirmed diagnosis of a solid tumor malignancy, excluding lymphoma
* Chemotherapy-naïve or previously treated with not more than 1 non-taxane-containing chemotherapy (Enrollment of patients with a history of prior taxane therapy in the adjuvant setting is allowed provided at least 6 months have passed since the conclusion of that therapy.)
* ECOG performance status of 0 or 1
* Adequate bone marrow, hepatic, and renal function
* At least 3 weeks and recovery from effects of prior surgery and anticancer therapy, with resolution of any toxicity to not more than Grade 1

Exclusion Criteria:

* Brain metastasis or leptomeningeal disease
* Second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which patient has been disease-free for 5 or more years)
* Known history of human immunodeficiency virus infection or hepatitis B or hepatitis C infection
* Recurrent diarrhea, defined as more than 3 episodes than is usual in any 24-hour period within the 30 days prior to enrollment in this study
* Significant medical disease other than cancer
* Neuropathy at least Grade 2
* Difficulty swallowing
* Malabsorptive disorder
* Need for other anticancer treatment while receiving study medication
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity. A washout period of at least 2 weeks is required prior to the first dose of study medication.
* Pregnancy or lactation
* History of hypersensitivity to tesetaxel, capecitabine, 5-fluorouracil, or any of their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 30 days following the last dose of study medication
  Percentage of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Schwartzberg, MD, FACP, Principal Investigator — The West Clinic
Locations (1):
- The West Clinic, Memphis, Tennessee, United States